CLINICAL TRIAL: NCT04089293
Title: Does the Contact Between the Deep Surface of the Supraspinatus Muscle Tendon and the Posterior Superior Labrum Physiological ?
Brief Title: The Postero-superior Contact and Rotator Cuff Lesion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7461
Record Dates: First submitted 2019-07-19; First posted 2019-09-13 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-07

CONDITIONS: GLENOID CAVITY
Keywords: GLENOID CAVITY; HUMERAL HEAD; SHOULDER JOINT; SUPRASPINATUS MUSCLE; LABRUM; ABER POSITION; SCAPULOHUMERAL; INTERNAL IMPINGEMENT; ABDUCTED POSITION; SCAPULOHUMERAL JOINT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The possibility of physiological contact between the deep surface of the tendon of the supraspinatus muscle and the labrum and/or posterior superior glenoidal rim during an armed movement of the arm (abduction and external rotation or ABER position) has been described for many years. The physiological hypotheses put forward to explain this contact are first of all that the intrinsic mobility of the scapulohumeral joint is limited by these 2 structures, that an anterior instability or micro-instability induces an abnormal anterior translation when performing an abduction and lateral rotation movement, or finally that there is a decrease in humeral retroversion. When this contact becomes symptomatic, it is called a posterior superior conflict. This pathology is mainly found in throwing athletes or athletes repeating maximum external rotation in the abducted position of the arm. This conflict is also described among some manual workers, and is then observed in an older age group.

ELIGIBILITY:
Inclusion criteria:

* Major subject ((≥18 years old)
* Operated subject (at the HUS between 01/01/2012 and 31/12/2013) under arthroscopy of anterior instability, of an unruptured tendinopathy of the rotator cuff, or of an extra-articular pathology.
* Subject not expressing opposition to the use of his data for research purposes

Exclusion criteria:

* Subject having expressed his opposition to participating in the study
* Patient under safeguard of justice
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated at the Hopitaux Universitaires de Strasbourg between 01/01/2012 and 31/12/2013 under arthroscopy of anterior instability, uninjured tendinopathy of the rotator cuff, or extra-articular pathology.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Study of posterior-superior contact in a patient with no rotator cuff lesion. | The period from January 1st, 2012 to December 31st, 2013 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CLAVERT, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de chirurgie du membre supérieur Hautepierre 2, Strasbourg, France